CLINICAL TRIAL: NCT06309108
Title: The Effect of Education Given to Patients With Two Different Materials Before Bariatric Surgery on Early Complications
Brief Title: Bariatric Surgery and Patient Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gülsüme Satir, Istanbul University- Cerrahpaşa PhD student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/68-04; İUC (Other: İUC)
Record Dates: First submitted 2023-12-15; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Bariatric Surgery Candidate; Education; Patient Education

STUDY DESIGN:
Intervention Model Description: In our study, patients who would undergo bariatric surgery were selected randomly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Education Group (Experimental): Education group was given training with a training booklet.
  Interventions: Other: Education Booklet
- Augmented Reality Group (Experimental): Augmented reality group was given training with a augmented reality with 3DQR application.
  Interventions: Other: Augmented Reality Group
- Control Group (No Intervention): Control group was given training with a hospital routine.

INTERVENTIONS:
Other: Education Booklet — The education group was given training with a education booklet
  Arms: Education Group
Other: Augmented Reality Group — The second of the intervention group was trained with augmented reality. Patients were able to see the augmented reality element with the 3DQR application.
  Arms: Augmented Reality Group

SUMMARY:
Obesity is a disease that poses a health risk and is increasing worldwide. Bariatric surgery is the most effective method used in the treatment of obesity. Preoperative health education for bariatric surgery patients is important to support surgery. There is not enough nursing research in the literature regarding training patients with two different materials before bariatric surgery. The purpose of the randomized controlled experimental study designed in light of this information was to determine the effect of education given to patients with two different materials before bariatric surgery on early complications. The rates of the study were determined by randomizing trial I, trial II, and control treatment in 66 rooms that met the interval and study screening criteria offered between May 2022 and June 2023 in the general surgery service of a university hospital. Data from the research; was collected with the Veria Total Form, Autar Risk Assessment Scale, Apfel Risk Score, Visual Comparison Scale-VAS (Visual Analog Scale-VAS), Training Satisfaction Survey, and Complication Monitoring Form. In the first face-to-face meeting in the experimental groups, we were given training by the researcher with the removable Training Booklet I and Training Booklet II and were monitored until discharge. No control group training was given.

DETAILED DESCRIPTION:
Training Booklet Group (Experimental Group I): Patients who were eligible for the research were informed about the purpose, content and method of the research by reading the volunteer information form, and verbal and written permission was obtained from those who agreed to participate in the research voluntarily. Before the surgery, Part I of the Data Collection Form and the Autar Risk Assessment Scale were recorded in the form by the researcher. Before the surgery, the patients were given Educational Booklet I. Patients' questions about the booklet were answered. The Education Satisfaction Survey was filled out by the patients in order to measure their satisfaction with the booklet. When the patient is taken to the service after the surgery, the Data Collection Form II. III. IV. Part V, Apfel Risk Score, VAS, and Complication Monitoring Form were evaluated and recorded until the patient was discharged.

Augmented Reality Group (Experiment II GROUP): Patients who were eligible for the research were informed about the purpose, content, and method of the research by reading the voluntary information form, and verbal and written permission was obtained from those who agreed to participate in the research voluntarily. Before the surgery, Part I of the Data Collection Form and the Autar Risk Assessment Scale were recorded in the form by the researcher. Before the surgery, the patients were given Educational Booklet II. They were asked to install the 3DQR Plus application on their smartphones. The patient's ability to scan the QR code was checked. Patients who could open and read the QR code and who could open 9 QR codes and see the augmented reality element were asked to fill out the Training Satisfaction Survey. When the patient is taken to the service after the surgery, the Data Collection Form II. III. IV. and Part V, Apfel Risk Score, VAS, and Complication Monitoring Form were evaluated and recorded until the patient was discharged.

Control Group Patients Patients who were eligible for the study were informed about the purpose, content, and method of the study by reading the voluntary information form.

Verbal and written permission was obtained from those who voluntarily agreed to participate in the study. Control group patients were not given any training by the researcher, and the service routine was applied. Before the surgery, Part I of the Data Collection Form and the Autar Risk Assessment Scale were recorded in the form by the researcher. When the patient is taken to the service after the surgery, the Data Collection Form II. III. IV. and Part V, Apfel Risk Score, VAS, and Complication Monitoring Form were evaluated and recorded until the patient was discharged.

ELIGIBILITY:
Inclusion Criteria:

* Able to use a smart phone with internet access
* Able to communicate visually and verbally,
* Individuals who can speak, understand and read Turkish are included in the research.

was done.

Exclusion Criteria:

* Unable to use the application,
* Those who want to leave the study for any reason,
* Patients who did not accept the study were not included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Veria Total Form for sociodemographic features | [Time Frame: 1 week]

SECONDARY OUTCOMES:
Autar Risk Assessment Scale for DVT | 1 week

OTHER OUTCOMES:
Apfel Risk Score for nausea and vomiting | 1 week
Visual Analog Scale-VAS for pain | 1 week
Training Satisfaction Survey | 1 week
Complication Monitoring Form to determine whether complications develop | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul University- Cerrahpasa Instutite Graduate Studies, Istanbul, Avcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No